CLINICAL TRIAL: NCT07319533
Title: Investigating the Effect of Exosome Derived From Human Fetal Umbilical Cord Mesanchymal Cells as Complimintary Treatment in Moderate to Severe Erectile Dysfunction
Brief Title: Clinical Trial Investigating the Effect of Exosomes as a Complementary Treatment in Severe to Moderate Erectile Dysfunction
Acronym: MSC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Labbafinejad Medical Center (Other)
Responsible Party: Principal Investigator, Amirhossein Kashi, Doctor Amirhossein Kashi, Labbafinejad Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SBMU.UNRC.REC.1403.015; IRCT20160406027253N3 (Other: IRCT (Iranian Registary ofClinical Trials))
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Erectile Dysfunction; Erectile Dysfunction Associated With Type 2 Diabetes Mellitus; Erectile Dysfunction Due to Arterial Disease; Erectile Dysfunction Due to Arterial Insufficiency; Erectile Dysfunction Due to General Medical Condition; Erectile Dysfunction Due to Neuropathy
Keywords: Erectile Dysfunction; Exosome; Mesanchymal Stem Cell; MSC
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A single blinded randomized clinical trail with a placebo-controlled group, consisting 70 patients in total (35 patients in each arm)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Exosome) (Experimental): patients in this arm will be injected 5 ml of exosome in corpus cavernosa of each side (2.5 ml in each side at base of the penis). This will happen once a week, for 6 weeks. Inorder to prevent the injected substance from spreading systemically, a tourniquet will be placed at the base of the penis for 10 minute following injection.
  Interventions: Biological: exosomes derived from human umbilical cord mesenchymal stem cells
- Control (Placebo Comparator): Control group: these patients will recieve 5 ml of intracavernosal normal saline (2.5 ml in each side of penile base). This will happen once a week, for 6 weeks. Inorder to prevent the injected substance from spreading systemically, a tourniquet will be placed at the base of the penis for 10 minute following injection.
  Interventions: Biological: Normal (0.9%) saline

INTERVENTIONS:
Biological: exosomes derived from human umbilical cord mesenchymal stem cells — Intervention group: patients in this group will be injected 5 ml of exosome in corpus cavernosa of each side (2.5 ml in each side at base of the penis). This will happen once a week, for 6 weeks. Inorder to prevent the injected substance from spreading systemically, a tourniquet will be placed at the base of the penis for 10 minute following injection.
  Arms: Intervention (Exosome)
Biological: Normal (0.9%) saline — Control group: these patients will recieve 5 ml of intracavernosal normal saline (2.5 ml in each side of penile base). This will happen once a week, for 6 weeks. Inorder to prevent the injected substance from spreading systemically, a tourniquet will be placed at the base of the penis for 10 minute following injection.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to Investigate the Effect of Injection of MSC-Derived Exosome on Patients with Erectile Dysfunction in overall healthy males, aged 18-70, with-out any severe active medical condition, with moderate to severe erectile dysfunction based on IIEF-5, and non-satisfactory response to other treatments (5PDEI). The main question it aims to answer is:

• Is MSC-derived exosome safe and effective in treating patients with ED by improving IIEF-5 score?

If there is a comparison group: Researchers will compare the intervention group (Exosome receiving group) with control group (placebo receiving group) to see if exosomes are safe and effective in treating male adult patients with moderate-sever ED.

Participants will receive six weekly injections of normal saline or exosome (based on group), and will undergo necessarily follow up, and examinations and observation.

DETAILED DESCRIPTION:
Secondary outcomes are the folllowing:

EHS score length of erected penis lenght of flacid penis (pulled) peak systolic volume (via dupler sonography) end diastolic volume (via dupler sonography) any adverse effects of exosome

ELIGIBILITY:
Inclusion Criteria:

Moderate or severe erectile dysfunction (according to IIEF-5) Non-satisfactory response to other treatments Generally Healthy males Not having severe past medical history

Exclusion Criteria:

Known allergy or history of hyperactivity to biological substances Peyronie's plaque Existing medical condition (severe or uncontrolled) Use of psychiatric medication Use of thyroid medication Hyopgonadism Hypergonadism Cancer History of prostatectomy Prostitis Autoimmune disease Recent trauma or surgery Ongoing systemic infection Skin lesion or infection at the site of injection

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
IIEF-5 score | week 0, 7, 13, 25, 49
  Erectile dysfunction of the patients during the study will be assessed by IIEF-5 questionnaire. It will done in a interview with the patients.

SECONDARY OUTCOMES:
EHS score | week 0, 7, 13, 25, 49
  Erectile Hardness Score It will be done in a interview with the patients.
Peak Systolic Voulme | week 0, 7, 13
  Peak systolic volum or arterial blood flow of the penis, which will be assessed by doppler sonography after papaverin injection
End Diastolic Volume | week 0, 7, 13
  end diastolic volume or venous blood flow of the penis which will be assessed by doppler sonography after papaverin injection
Pulled length of penis | week 0, 7, 13, 25, 49
  the pulled length of penis which will be assessed by clinician at each follow up session
Erected length of Penis | week 0, 7, 13, 25, 49
  erected length of penis which will be assessed at follow up sessions by clinician
Side effects | week 1, 2, 3, 4, 5, 6
  any immeadiate, or late onset local side effects at injection site. these will be reported both by the patients and assessed by the clinician.

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Labbafinejad Hospital, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make this available.